CLINICAL TRIAL: NCT05948748
Title: Preoperative Anxiety Level and Associated Factors in Patients Undergoing Minimally Invasive Osteoarticular Foot Surgery
Brief Title: Level of Anxiety in Patients Undergoing Invasive Foot Surgery
Status: Completed | Type: Observational
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal investigator, Universidad Católica de Ávila
Other Study IDs: 08/07/2023
Record Dates: First submitted 2023-07-08; First posted 2023-07-17 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Anxiety Postoperative; Surgery
Keywords: anxiety; surgery; minor surgical procedures; postoperative pain
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anxiety levels: pre-surgical anxiety levels in patients undergoing minimally invasive osteoarticular foot surgery
  Interventions: Procedure: foot surgery

INTERVENTIONS:
Procedure: foot surgery — minimally invasive osteoarticular foot surgery

SUMMARY:
In recent decades, preoperative anxiety has been studied by numerous authors from different medical-surgical specialties, however, there are no studies in the scientific literature on anxiety prior to surgical procedures in the area of minimally invasive foot surgery at the osteoarticular level.

The aim of the present study was to determine the level of preoperative anxiety and information using the Amsterdam Preoperative Anxiety and Information scale in patients undergoing minimally invasive podiatric surgery, as well as to determine the socio-demographic and surgical factors associated with preoperative anxiety.

ELIGIBILITY:
Inclusion Criteria:

* be over18 years old.
* ASA I and II (American Society of Anesthesiologists).
* autonomous capacity to fill out the surveys and participate in the study

Exclusion Criteria:

* mental and/or emotional disorders.
* incapacity to understand.
* people medicated with anxiolytics before the surgery.
* chronic pain in the foot and/or analgesic treatment for chronic pain.
* did not fulfill the postoperative recommendations.
* contraindication to the study's medical guideline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing minimally invasive osteoarticular foot surgery
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
pre-surgical anxiety levels | 1 day
  Amsterdam Pre-Operative Anxiety and Information Scale (APAIS) using a 5-point Likert scale, where 1 = not at all and 5 = total.

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge V Velázquez Saornil, Ávila, Avila, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laufenberg-Feldmann R, Kappis B, Schuster M, Ferner M. [Relevance of preoperative anxiety for postoperative outcome in urological surgery patients: A prospective observational study]. Schmerz. 2016 Apr;30(2):166-73. doi: 10.1007/s00482-015-0023-3. German. PMID 26242358
- [Background] Guo P, East L, Arthur A. A preoperative education intervention to reduce anxiety and improve recovery among Chinese cardiac patients: a randomized controlled trial. Int J Nurs Stud. 2012 Feb;49(2):129-37. doi: 10.1016/j.ijnurstu.2011.08.008. Epub 2011 Sep 22. PMID 21943828
- [Background] Navarro-Garcia MA, Marin-Fernandez B, de Carlos-Alegre V, Martinez-Oroz A, Martorell-Gurucharri A, Ordonez-Ortigosa E, Prieto-Guembe P, Sorbet-Amostegui MR, Indurain-Fernandez S, Elizondo-Sotro A, Irigoyen-Aristorena MI, Garcia-Aizpun Y. [Preoperative mood disorders in patients undergoing cardiac surgery: risk factors and postoperative morbidity in the intensive care unit]. Rev Esp Cardiol. 2011 Nov;64(11):1005-10. doi: 10.1016/j.recesp.2011.06.009. Epub 2011 Sep 15. Spanish. PMID 21924811
- [Result] Navarro-Gaston D, Munuera-Martinez PV. Prevalence of Preoperative Anxiety and Its Relationship with Postoperative Pain in Foot Nail Surgery: A Cross-Sectional Study. Int J Environ Res Public Health. 2020 Jun 22;17(12):4481. doi: 10.3390/ijerph17124481. PMID 32580413
- [Result] Zelenikova R, Homzova P, Homza M, Buzgova R. Validity and Reliability of the Czech Version of the Amsterdam Preoperative Anxiety and Information Scale (APAIS). J Perianesth Nurs. 2017 Oct;32(5):429-437. doi: 10.1016/j.jopan.2016.03.007. Epub 2016 Dec 28. PMID 28938978
- [Result] Wu H, Zhao X, Chu S, Xu F, Song J, Ma Z, Gu X. Validation of the Chinese version of the Amsterdam Preoperative Anxiety and Information Scale (APAIS). Health Qual Life Outcomes. 2020 Mar 11;18(1):66. doi: 10.1186/s12955-020-01294-3. PMID 32160883
- [Result] Aust H, Eberhart L, Sturm T, Schuster M, Nestoriuc Y, Brehm F, Rusch D. A cross-sectional study on preoperative anxiety in adults. J Psychosom Res. 2018 Aug;111:133-139. doi: 10.1016/j.jpsychores.2018.05.012. Epub 2018 May 22. PMID 29935747
- [Result] Vergara-Romero M, Morales-Asencio JM, Morales-Fernandez A, Canca-Sanchez JC, Rivas-Ruiz F, Reinaldo-Lapuerta JA. Validation of the Spanish version of the Amsterdam Preoperative Anxiety and Information Scale (APAIS). Health Qual Life Outcomes. 2017 Jun 7;15(1):120. doi: 10.1186/s12955-017-0695-8. PMID 28592310